CLINICAL TRIAL: NCT07384429
Title: Study for the Dual Orexin Receptor Antagonist Lemborexant in Improving Motor-Sleep Comorbidity in Parkinson's Disease
Brief Title: Effects of Lemborexant on Motor-sleep Comorbidity in Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: YangPan (Other)
Collaborators: Eisai China Inc. (Industry); Nanjing University (Other)
Responsible Party: Sponsor-Investigator, YangPan, Chief Physician, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025401
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease; Insomnia; Motor Disorder
Keywords: Parkinson's Disease; Lemborexant; orexin receptor antagonist; Insomnia; Motor Disorder
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders; Motor Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): oral matching placebo
  Interventions: Drug: placebo
- Lemborexant (Experimental): oral Lemborexant (5 mg/day)
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — Participants will receive oral Lemborexant (5 mg/day) nightly approximately 5-30 minutes before going to bed for 28 consecutive days.
  Arms: Lemborexant
Drug: placebo — Participants will receive a matching placebo nightly approximately 5-30 minutes before going to bed for 28 consecutive days.
  Arms: placebo

SUMMARY:
The aim of this study is to explore the effects of the dual orexin receptor antagonist Lemborexant on improving motor and sleep comorbidity in patients with Parkinson's disease. This study will provide clinical evidence for the application of dual orexin receptor antagonists in the treatment of Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the most common movement disorder. Its core motor symptoms include bradykinesia, resting tremor, muscle rigidity, and postural instability. Furthermore, patients frequently experience severe non-motor symptoms, such as sleep disorders and mood/affective disturbances. Among these, sleep disorders, especially insomnia, are one of the most prevalent non-motor symptoms. They are often overlooked in clinical management. The axons of central orexin neurons project extensively throughout the brain, encompassing key regions such as motor control centers and sleep-wake regulation centers. During the pathological process of PD, dysfunctional orexin neurons may contribute to the disruption of both motor and sleep functions by modulating these target areas.

By recruiting PD patients with comorbid motor and insomnia symptoms, the investigators will investigate the efficacy of Lemborexant in treating both motor and sleep disturbances in PD patients. With its advantages of target specificity, established safety, and a lower side-effect profile compared to traditional hypnotics, Lemborexant holds promise as a novel therapeutic intervention for Parkinson's disease. This research may offer new possibilities for expanding clinical treatment strategies for PD. Participants will take 5 mg medication (or placebo) each night for 28 days and be asked to come for 4 times study visits (Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up).

The major experiment contents include:

1. To evaluate the effect of oral Lemborexant on Parkinson's disease motor symptoms in participants (using the Unified Parkinson's Disease Rating Scale, UPDRS);
2. To evaluate the effect of oral Lemborexant on the sleep quality of participants (using the Parkinson's Disease Sleep Scale (PDSS), the Insomnia Severity Index (ISI), the Pittsburgh Sleep Quality Index (PSQI)).

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 50 years or older;
* 2. Diagnosed with idiopathic Parkinson's disease according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease (2015), with a Hoehn & Yahr stage of 1 to 4;
* 3. Disease duration of ≥ 2 years since diagnosis, clinically stable, and able to comply with the research assessments and interventions;
* 4. Diagnosis of insomnia disorder meeting the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with an Insomnia Severity Index (ISI) score of ≥ 15;
* 5. Stable medication regimen for at least 4 weeks prior to the study;
* 6. Signed informed consent form, with the participant or their legal guardian able to understand and willing to participate in this study.

Exclusion Criteria:

* 1. History of or diagnosis with a severe psychiatric disorder, such as depression, anxiety disorders, schizophrenia spectrum disorders, or bipolar disorder;
* 2. Presence of a clinically defined neurological disorder (assessed via self-report), including but not limited to: any condition potentially associated with increased intracranial pressure, space-occupying brain lesions, history of stroke, transient ischemic attack within the past 2 years, cerebral aneurysm, dementia, or multiple sclerosis;
* 3. Severe cognitive impairment (Mini-Mental State Examination (MMSE) score below 24) or inability to complete questionnaires independently;
* 4. Chronic obstructive pulmonary disease (COPD) or any lifelong history of sleep-related breathing disorders, such as sleep apnea;
* 5. Excessive daytime sleepiness, defined as self-reported daily daytime napping ≥ 1 hour per day on ≥ 3 days per week;
* 6. Regular caffeine consumption;
* 7. Use of any orexin receptor related medication within the past 3 months.
* 8. Previous history of cataplexy or known reduced orexin levels;
* 9. Inability to read or understand Chinese;
* 10. Use of other sleep-promoting medications within the past 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the scores of Part III of the Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up.
  The scores of Part III of the UPDRS (motor examination) score will be collected from each participant to measure the severity of motor ability with scores ranging from 0 (minimum) to 108 (maximum). The higher scores mean a worse outcome.
Changes in the scores of the Parkinson's Disease Sleep Scale (PDSS) | Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up.
  PDSS is used to quantify the severity of sleep problems associated with Parkinson's disease. Its score ranges from 0 (minimum) to 150 (maximum), with lower scores indicating more severe sleep disturbances. Typically, a total score below 90 is considered indicative of a clinically significant sleep disorder.

SECONDARY OUTCOMES:
Changes in the scores of Part II of the Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up.
  The scores of Part II of the UPDRS (daily living activities) score will be collected from each participant to measure the severity of daily living activities with scores ranging from 0 (minimum) to 52 (maximum). The higher scores mean a worse outcome.
Changes in the scores of the Insomnia Severity Index (ISI) | Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up.
  ISI is used to screen for and assess the severity of insomnia. Its score ranges from 0 (minimum) to 28 (maximum), with higher scores indicating more severe sleep problems. A total score of 10 or above suggests the presence of clinically significant insomnia.
Changes in the scores of the Pittsburgh Sleep Quality Index (PSQI) | Baseline, at the end of the 7-day post-treatment, at the end of the 28-day post-treatment, 7-day follow up.
  PSQI is used to comprehensively evaluate multiple aspects of sleep quality. Its score ranges from 0 (minimum) to 21 (maximum), with higher scores indicating poorer sleep quality. A total score greater than 5 is generally considered to indicate poor sleep quality.